CLINICAL TRIAL: NCT00427596
Title: A Two-Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Four MR Formulations and Food Effect of GW427353 (Solabegron) in Healthy Adult Subjects
Brief Title: A Two-Part Study to Determine: Best Medication Formulation and Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3A106044
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Overactive Bladder
Keywords: GW427353 oral tablets,; healthy adult subjects,; food effect
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — solabegron

INTERVENTIONS:
Drug: Solabegron

SUMMARY:
This is a two-part study. Part 1 is designed to find the best modified release formulation of GW423753; Part 2 is designed to use the selected formulation(s) from Part 1 to find out if food affects the way the medication is processed by the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males & females
* Part 1 ages 18-60
* Part 2 ages 18-50 & 65-80
* Within normal weight range given your height
* Negative urine drug and alcohol test
* Willing to follow all study procedures

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening physical examination, clinical laboratory tests, 12-lead ECG, or any other medical condition or circumstance making the subject unsuitable for participation in the study based on the Investigator's assessment.
* Subjects with either a blood pressure measurement > 150/90 mmHg, or a history of coronary disease AND a blood pressure > 140/90 mmHg, at screening.
* History of drug or other allergy, which, in the opinion of the Investigator, contraindicates their participation.
* Regular alcohol consumption averaging >/7 drinks/week for women or >/ 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of the first dose of study medication.
* Positive urine drug, alcohol or serum pregnancy test at screening and prior to dosing in each study session.
* Positive for hepatitis C antibody, hepatitis B surface antigen or HIV at screening.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to administration of study medication.
* Use of prescription or non-prescription drugs within 7 days or 5 half-lives (whichever is longer) prior to administration of study medication and during the study. By exception, use of acetaminophen at doses of ≤ 2 grams per day, the use of contraceptives (oral, depots, patches, etc.) and anti-hypertensive medications will be permitted.
* Use of vitamins or herbal/dietary supplements within 7 days prior to administration of study medication and during the study.
* Subject is unable and/or unwilling to adhere to Lifestyle Guidelines
* Subjects who have donated more than 500 mL of blood or plasma within 56 days prior to administration of study medication.
* An unwillingness on the part of male volunteers to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness to use a condom and another form of contraception (e.g., IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant from the time of the first dose of study medication until completion of follow-up procedures.
* Pregnant or lactating woman. A pregnancy test will be performed for all women at screening and prior to each dosing session to confirm eligibility.
* The subject has a known hypersensitivity or idiosyncratic reaction to any drug chemical related to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Absorption rate of the tablet formulations as measured several times by blood draws (over 48-hour period) during the Part 1 under fed conditions and Part 2 under fed vs. fasted conditions

SECONDARY OUTCOMES:
Toleration of the formulations after single and repeat doses (over 7-day period)
Part 1: Safety and tolerability assessments will include data from spontaneous adverse event reporting, vital signs, 12-lead ECGs, physical examinations, and safety laboratory tests.
Part 2: Safety and tolerability assessments will include data from spontaneous adverse event reporting, vital signs, 12-lead ECGs, physical examinations, and safety laboratory tests.
Part 2: The secondary pharmacokinetic parameters will be the AUC, Cmax, Tmax, and T1/2 following repeat oral dosing of Solabegron, as the data permit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, MSc, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States